CLINICAL TRIAL: NCT04210726
Title: Effect of Human Body Immersion in Hypertonic Saline Solution on Cancer Nodules' Size, Number and Its Metastasis Properties in Vivo.
Brief Title: Effect of Salt Solution Immersion Bath on Cancer in Vivo.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Working on complying with the Research Ethics Board requirements.
Sponsor: Rafik Batroussy (Other)
Responsible Party: Sponsor-Investigator, Rafik Batroussy, Principal Investigator, Batroussy, Rafik
Organization: Batroussy, Rafik (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-12-21; First posted 2019-12-26 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A pilot randomized blinded controlled study, whereas a number of patients with clinically-diagnosed Cancer (any type, any location and any stage), and who were poorly responsive to at least one cycle of conventional and standard therapy (Chemotherapy or Radiation therapy), are equally divided into 2 groups, Active and Control groups. The Active group patients will separately have an immersion bath in 25% Sea Salt in Water solution at a temperature comfortable to every patient, whereas the bath solution is in direct contact with the skin, for 30 minutes once daily for 7 consecutive days, in addition to their standard treatments they receive from their health care providers. The Control group's patients will separately have a bath in 0.9% Sea Salt in Water at a comfortable temperature whereas the bath solution is in direct contact with the skin, for 30 minutes once daily for 7 consecutive days, in addition to their standard treatments they receive from their health care providers.
Who Masked: Participant
Masking Description: Participants will not know which Group (Active/Control) they are assigned to, only the Investigator will know. The amount of Salt added to each bath (and hence the concentration of each bath) will not be known by Participants. Assignment will be random using a simple computer program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group - 25% Saline Bath (Active Comparator): The Active group's patients will separately have an immersion bath in 25% Sea Salt in Water solution (made by adding pure Sodium Chloride in the form of Sea Salt to Tap Water Bath) at a temperature comfortable to every participant (please note that Solubility of Sodium Chloride in Water does not change significantly with change in temperature, therefore the concentration will remain the same regardless of water temperature), whereas the bath solution is in direct contact with the skin, for 30 minutes once daily for 7 consecutive days, in addition to their standard treatments they receive from their health care providers.
  Interventions: Drug: 25% Hypertonic Saline Bath
- Control Group - 0.9% Saline Bath (Placebo Comparator): The Control group's patients will separately have a bath in 0.9% Sea Salt in Water (Isotonic solution, made by adding Sodium Chloride in form of Sea Salt to Tap Water) at a comfortable temperature whereas the bath solution is in direct contact with the skin, for 30 minutes once daily for 7 consecutive days, in addition to their standard treatments they receive from their health care providers
  Interventions: Other: 0.9% Isotonic Saline Bath

INTERVENTIONS:
Drug: 25% Hypertonic Saline Bath — 25% Sea Salt (mainly Sodium Chloride - NaCl) in Tap Water Immersion Bath (made by adding Sodium Chloride in the form of Sea Salt to Tap Water to a concentration of 25%).
  Arms: Active Group - 25% Saline Bath
Other: 0.9% Isotonic Saline Bath — 0.9% Sea Salt (mainly Sodium Chloride - NaCl) in Tap Water Immersion Bath (made by adding Sodium Chloride in the form of Sea Salt to Tap Water to a concentration of 0.9%).
  Arms: Control Group - 0.9% Saline Bath

SUMMARY:
This Study evaluates the effectiveness of Hypertonic Saline Bath in reducing the Cancer nodules' size, number and SUVmax.

DETAILED DESCRIPTION:
Many previous studies have shown that the Cancer cells are over-hydrated, and that Hyponatraemia exists in many cases of Cancer. The Cancer cell's viability depends on Angiogenesis and formation of blood vessels that carry water and nutrient to the rapidly-dividing Cancer cells. This study tests the hypothesis that disrupting the water content of blood could lead to increasing its Tonicity and hence withdrawing water from the Cancer cells by Osmosis, which can result in disrupting the growth of the Cancer cell itself. This disruption of Blood Water content can be achieved using Osmotic Pressure differential via immersing the whole body in Hypertonic Saline Solution for a certain amount of time, thus making the Blood more Hypertonic relative to the cells of the body and of the cancer, leading to water withdrawal from the cells of the body and of the cancer. While body's cells can sustain temporary dehydration, Cancer cells could be negatively affected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PET/CT scan-confirmed Cancer (any type, any location and any stage) who have poorly responded to at least one cycle of conventional and standard therapy (Chemotherapy, Radiation or Drug therapy) .
* Age 5 to 80 years old
* Life expectancy of at least 1 year
* Can understand and read English
* Lives in Calgary Alberta

Exclusion Criteria:

Patients with the following medical conditions will be excluded:

1. Kidney diseases
2. Dialysis
3. Fever
4. On Blood Thinners or with any Coagulation disorder
5. History of stroke
6. Hypernatraemia
7. Hypotension (Low Blood Pressure)
8. Hypovolemia/Dehydration
9. Tachycardia (Rapid Heart rate)
10. Epilepsy
11. Open wounds
12. Any medical condition that might cause the patient to lose consciousness
13. Participants who cannot tolerate thirst during the 30 minutes bath.
14. Participants who are not residents of Calgary Alberta Canada with a valid Alberta Health Card.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in Tumors size | 6 month
  Tumor responses are evaluated in terms of change in tumor size represented by the linear measurements of all targeted lesions. The Hypertonic Sea Salt Bath intervention will be considered effective if there is a statistically-significant reduction in Means of the measured Cancer Cells sizes/dimensions for the same nodules between the two groups using a One-Way ANOVA test.
Reduction in Tumors lesions numbers | 6 month
  Tumor responses are evaluated in terms of change in tumor lesions number. The Hypertonic Sea Salt Bath intervention will be considered effective if there is a statistically-significant reduction in Means of the Cancer lesions number for the same nodules between the two groups using a One-Way ANOVA test.
Reduction in Tumors lesions SUVmax (FDG-Maximum Standardized Uptake Values) | 6 month
  Tumor responses are evaluated in terms of change in tumor SUV max (FDG-Maximum Standardized Uptake Values). The Hypertonic Sea Salt Bath intervention will be considered effective if there is a statistically-significant reduction in Means of the measured Cancer lesions SUVmax values for the same nodules between the two groups using a One-Way ANOVA test.

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Batroussy, Study Chair — Independent Researcher
Locations (1):
- Rafik Batroussy, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntyre GI. Cell hydration as the primary factor in carcinogenesis: A unifying concept. Med Hypotheses. 2006;66(3):518-26. doi: 10.1016/j.mehy.2005.09.022. Epub 2005 Nov 3. PMID 16271440
- [Background] Machado M, Salgado TM, Hadgraft J, Lane ME. The relationship between transepidermal water loss and skin permeability. Int J Pharm. 2010 Jan 15;384(1-2):73-7. doi: 10.1016/j.ijpharm.2009.09.044. Epub 2009 Sep 30. PMID 19799976
- See also: Synthetic ion transporters can induce apoptosis by facilitating chloride anion transport into cells. — https://www.nature.com/articles/nchem.2021
- See also: High Salt Inhibits Tumor Growth by Enhancing Anti-tumor Immunity. — https://www.frontiersin.org/articles/10.3389/fimmu.2019.01141/full
- See also: Cell swelling, softening and invasion in a three-dimensional breast cancer model. — https://www.nature.com/articles/s41567-019-0680-8
- See also: Cell Stiffness May Indicate Likelihood of Cancer Metastasis. — https://www.genengnews.com/news/cell-stiffness-may-indicate-likelihood-of-cancer-metastasis/
- See also: The Dysfunction of Metabolic Controlling of Cell Hydration Precedes Warburg Phenomenon in Carcinogenesis — https://www.longdom.org/open-access/the-dysfunction-of-metabolic-controlling-of-cell-hydration-precedes-warburg-phenomenon-in-carcinogenesis-jbb.10000e59.pdf